CLINICAL TRIAL: NCT05585528
Title: Effect of Informing the Patient on the Type of Management, Surgical or Functional, After Rupture of the Anterior Cruciate Ligament : INFO-LCA
Brief Title: Informing the Patient on the Type of Management, Surgical or Functional, After Rupture of the Anterior Cruciate Ligament
Acronym: INFO-LCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-A00931-42
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Ligament Rupture
MeSH Terms: interventions — Functional Status

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal, open, non-comparative (single arm), monocentric study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type of management, surgical or functional, after rupture of the anterior cruciate ligament (Other): Patients will choose the type of management, surgical or functional, after rupture of the anterior cruciate ligament.
  Interventions: Procedure: Functional or surgical management in 1st intention

INTERVENTIONS:
Procedure: Functional or surgical management in 1st intention — Proportion of patients after rupture of the anterior cruciate ligament of the knee, who will have functional or surgical management in 1st intention

SUMMARY:
The purpose of the study is to evaluate the proportion of patients after rupture of the anterior cruciate ligament (ACL) of the knee, who will have functional or surgical management (PEC) in 1st intention, after having received appropriate information.

DETAILED DESCRIPTION:
As part of this study, patients will be followed for 1 year with regular functional and quality of life assessments (45 days after inclusion, 3, 6, 9 and 12 months after the start of surgical or non-surgical management). Patients who, during follow-up, will have been redirected towards surgery by the doctor (in the event of functional instability) or who will have chosen to finally move towards surgical PEC, will also be followed.

ELIGIBILITY:
Inclusion Criteria:

* Rupture, partial or complete, of the anterior cruciate ligament less than 3 months old (confirmed by magnetic resonance imaging);
* Patient with no contraindication to surgery or functional management, according to the medical team;
* Patient able to understand the information related to the study, to read the information leaflet and having consented to participate in the study
* Patient benefiting from a social security scheme;

Exclusion Criteria:

* Grade 3 associated ligament injury on the fibular collateral ligament and/or the tibial collateral ligament;
* Symptomatic meniscal lesion;
* Practice of sport in national or international competition ;
* Recurrence of rupture of the same anterior cruciate ligament;
* Patient with a neurological (motor and/or sensory), vestibular or rheumatic pathology;
* Pregnant woman ;
* Protected adult patient (under guardianship, or under a regime of deprivation of liberty).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients operated at 45 days | 45 days
  Rate of patients in the total population who underwent surgery 45 days after anterior cruciate ligament rupture

SECONDARY OUTCOMES:
Proportion of patients who persist in the choice of non-surgical | 12 months
  To assess the proportion of patients who persist in the choice of non-surgical management at 3, 6, 9 and 12 months (in patients who had initial non-surgical management).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No